CLINICAL TRIAL: NCT04670601
Title: Bioequivalence Study of Flurbiprofen 8.75 mg Lozenge vs. the Reference Product Strepfen 8.75 mg Lozenge in Healthy Volunteers
Brief Title: Bioequivalence of Flurbiprofen Lozenge vs Strepfen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 073WO18070; CRO-PK-18-329 (Other: CROSS Research)
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: flurbiprofen; lozenge; Strepfen; bioequivalence
MeSH Terms: interventions — strepfen

STUDY DESIGN:
Intervention Model Description: Single dose, open-label, randomised, 2-way cross-over bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flurbiprofen 8.75 mg (Experimental): Flurbiprofen 8.75 mg lemon and honey flavour lozenge
  Interventions: Drug: Flurbiprofen Test 8.75 MG
- Strepfen 8.75 mg (Active Comparator): Strepfen 8.75 mg lemon and honey lozenge
  Interventions: Drug: Flurbiprofen Reference 8.75 MG

INTERVENTIONS:
Drug: Flurbiprofen Test 8.75 MG — Subjects will be asked to swallow saliva before dosing. For each administration, subjects will move the lozenge around in their mouth, suck on the lozenge continually for 15 min and swallow saliva at any time during the product administration procedures, being very careful not to swallow the lozenge.
  Arms: Flurbiprofen 8.75 mg
Drug: Flurbiprofen Reference 8.75 MG — Subjects will be asked to swallow saliva before dosing. For each administration, subjects will move the lozenge around in their mouth, suck on the lozenge continually for 15 min and swallow saliva at any time during the product administration procedures, being very careful not to swallow the lozenge.
  Other Names: Strepfen
  Arms: Strepfen 8.75 mg

SUMMARY:
The present study has been designed to compare flurbiprofen pharmacokinetic profile after administration of flurbiprofen 8.75 mg lozenges, marketed by ACRAF, S.p.A., Italy (test product), and the marketed Strepfen 8.75 mg honey and lemon lozenges reference product. (Reckitt Benckiser Portugal SA).

DETAILED DESCRIPTION:
This is a single dose, open-label, randomised, 2-way cross-over bioequivalence study aimed to compare the bioavailability and the plasma pharmacokinetic profile of flurbiprofen after single dose administration of test and reference formulations.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: signed written informed consent before inclusion in the study.
* Sex and Age: males and females, 18-55 years old inclusive.
* Habits: non smokers.
* Body Mass Index (BMI): 18.5-30 kg/m2 inclusive.
* Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, heart rate (HR) 50-90 bpm, measured after 5 min at rest in the sitting position.
* Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study.
* Contraception and fertility (women only): females of child-bearing potential must be using at least one of the following reliable methods of contraception:
* Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
* A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
* A male sexual partner who agrees to use a male condom with spermicide
* A sterile sexual partner Women of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted.

For all women, pregnancy test result must be negative at screening and day -1.

Exclusion Criteria:

* Electrocardiogram (12-lead ECG in supine position): clinically significant abnormalities.
* Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study; subjects with dry mouth conditions or with any other diseases/problems of the mouth which the investigator considers may affect the outcome of the study.
* Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness.
* Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study.
* Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study.
* Medications: medications, including over the counter (OTC) medications and herbal remedies, in particular flurbiprofen, for 2 weeks before the start of the study. Hormonal contraceptives for females will be allowed
* Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
* Blood donation: blood donations for 3 months before this study
* Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2015-2020 (9)], or caffeine abuse (>5 cups coffee/tea/day); smokers
* Drug test: positive result at the drug test at screening or day-1
* Alcohol test: positive alcohol breath test at day -1
* Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
* Pregnancy (women only): positive or missing pregnancy test at screening or day -1, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration | pre-dose (0), 10, 20, 30, 40, 50 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  to evaluate the rate (Cmax) of absorption of flurbiprofen in plasma after single dose administration
Area under the plasma concentration-time curve 0-t | pre-dose (0), 10, 20, 30, 40, 50 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  to evaluate the extent of absorption of flurbiprofen in plasma after single dose administration

SECONDARY OUTCOMES:
Time to achieve Cmax | pre-dose (0), 10, 20, 30, 40, 50 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  to evaluate time to achieve Cmax
tlag | pre-dose (0), 10, 20, 30, 40, 50 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  to evaluate time prior to the first measurable (i.e. above lower quantification limit) concentration
Relative bioavailability of flurbiprofen in plasma | pre-dose (0), 10, 20, 30, 40, 50 minutes and 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours post-dose
  to evaluate relative bioavailability of flurbiprofen in plasma
Palatability | 2 times through the two week study period
  to assess the palatability of test and reference formulations using a 0-100 mm VAS where 0 mm indicated "not pleasant at all" and 100 mm indicated "very pleasant".
Treatment-Emergent Advers Events | through the two week study period
  to evaluate number of TEAEs and number of subjects with TEAEs

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — Cross Research S.A.
Locations (1):
- CROSS Research S.A., Phase I Unit, Arzo, Switzerland